CLINICAL TRIAL: NCT01521767
Title: A Single-Dose Pharmacokinetics And Relative Bioavailability Study Of Tolterodine From Two Microspheres In Powder Blend Extended Release Formulations Compared To The Commercial Extended Release Capsules
Brief Title: Pharmacokinetics and Relative Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A6121196
Record Dates: First submitted 2012-01-17; First posted 2012-01-31 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Urinary Bladder, Overactive
Keywords: pharmacokinetics; relative bioavailability; tolterodine microspheres in powder blend; Overactive Urinary Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Tolterodine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- A (Experimental): 4 mg tolterodine extended release capsules, administered with water and under fasting condition.
  Interventions: Drug: tolterodine tartrate
- B (Experimental): 4 mg microspheres in powder blend release rate 2 (MPB-RR2), administered without water and under fasting condition.
  Interventions: Drug: tolterodine tartrate
- C (Experimental): 4 mg microspheres in powder blend release rate 1 (MPB-RR1), administered without water and under fasting condition.
  Interventions: Drug: tolterodine tartrate
- D (Experimental): 4 mg MPB-RR1, administered without water and under fed condition.
  Interventions: Drug: tolterodine tartrate
- E (Experimental): 4 mg MPB-RR1, administered with water and under fasting condition.
  Interventions: Drug: tolterodine tartrate

INTERVENTIONS:
Drug: tolterodine tartrate — 4 mg single dose of extended release capsules
  Arms: A
Drug: tolterodine tartrate — 4 mg single dose of microspheres in powder blend
  Arms: B
Drug: tolterodine tartrate — 4 mg single dose of microspheres in powder blend
  Arms: C
Drug: tolterodine tartrate — 4 mg single dose of microspheres in powder blend
  Arms: D
Drug: tolterodine tartrate — 4 mg single dose of microspheres in powder blend
  Arms: E

SUMMARY:
A Single-Dose Pharmacokinetics And Relative Bioavailability Study Of Tolterodine From Two Microspheres In Powder Blend Extended Release Formulations Compared To The Commercial Extended Release Capsules

DETAILED DESCRIPTION:
Pharmacokinetics And Relative Bioavailability Study Of Tolterodine From Two Microspheres In Powder Blend Extended Release Formulations Compared To The Commercial Extended Release Capsules

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 21 and 55 years, inclusive

Exclusion Criteria:

* Evidence or history of clinically significant diseases

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of tolterodine | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 30, 36 hours post-dose
Maximum Observed Plasma Concentration (Cmax) of tolterodine | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 30, 36 hours post-dose

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of tolterodine. | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 30, 36 hours post-dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of 5-HMT | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 30, 36 hours post-dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of 5-HMT | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 30, 36 hours post-dose
Maximum Observed Plasma Concentration (Cmax) of 5-HMT | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 30, 36 hours post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) of tolterodine | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 30, 36 hours post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) of 5-HMT | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 30, 36 hours post-dose
Plasma Decay Half-Life (t1/2) of tolterodine | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 30, 36 hours post-dose
Plasma Decay Half-Life (t1/2) of 5-HMT | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 30, 36 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6121196&StudyName=Pharmacokinetics%20and%20Relative%20Bioavailability%20Study%20